CLINICAL TRIAL: NCT01868425
Title: ACL Repair and Multimodal Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-0538; 2017-0712 (Other: IRB ID); A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2013-05-13; First posted 2013-06-04 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Gabapentin; Ketamine; Bupivacaine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- multimodal:acetaminophen, gabapentin, ketamine, bupivacaine (Experimental): aggressive multimodal plus standard care, which includes ketorolac, bupivacaine, fentanyl, ondansetron, dexamethasone, sevoflurane
  Interventions: Drug: multimodal:acetaminophen, gabapentin, ketamine, bupivacaine
- placebo pills and injectables (Placebo Comparator): standard care which includes ketorolac, bupivacaine, fentanyl, ondansetron, dexamethasone, sevoflurane
  Interventions: Drug: placebo pills and injectables

INTERVENTIONS:
Drug: multimodal:acetaminophen, gabapentin, ketamine, bupivacaine — acetaminophen, gabapentin, ketamine, bupivacaine and standard care which includes ketorolac, bupivacaine, fentanyl, ondansetron, dexamethasone, sevoflurane
  Arms: multimodal:acetaminophen, gabapentin, ketamine, bupivacaine
Drug: placebo pills and injectables — receives standard care which includes ketorolac, bupivacaine, fentanyl, ondansetron, dexamethasone, sevoflurane plus placebos of intervention arm meds
  Arms: placebo pills and injectables

SUMMARY:
This study will evaluate the effectiveness of an aggressive multimodal regimen versus standard multimodal for Anterior Cruciate Ligament (ACL) repair using hamstring graft for patients having surgery in our outpatient surgicenter.

ELIGIBILITY:
Inclusion Criteria:

* Patients of orthopedic surgeons on the study team scheduled for ACL repair using hamstring graft from the same leg will be considered for inclusion in this study. Other inclusion criteria are as follows:

  * American Society of Anesthesiologists (ASA) physical status 1-3
  * BMI of < 40 kg/m2
  * Consents to general anesthesia and pre-operative femoral nerve block for case

Exclusion Criteria:

* Any contraindication to a femoral nerve block
* Allergy to local anesthetics, nonsteroidal anti-inflammatory medications, ketamine, acetaminophen, hydromorphone, oxycodone
* Peripheral or central nervous system disease
* Renal or hepatic impairment
* History of opioid dependence or current regular narcotic use
* Significant psychiatric disease
* Pregnancy or lactation (by verbal report)
* Seizure Disorder
* History of post-operative nausea and vomiting
* Latex allergy
* Clinically significant cardiac or pulmonary disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Shepler, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Started | 55 | 57
Completed | 55 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.5) | 32.2 (8.8) | 31.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 39 | 36 | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55 | 57 | 112
Smoking [Count of Participants; unit: Participants]
  Current Smoker | 3 | 9 | 12
  Former Smoker | 5 | 5 | 10
  Never a Smoker | 49 | 41 | 90
Weight [Mean (Standard Deviation); unit: kg] | 81.1 (15.8) | 82.2 (16.9) | 81.7 (16.3)
Height [Mean (Standard Deviation); unit: cm] | 175.9 (8.6) | 175.8 (8.6) | 175.9 (8.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.4) | 26.5 (4.3) | 26.4 (4.2)
ASA Physical Status [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA): ASA 1 - A normal healthy patient; ASA 2 - A patient with mild systemic disease
  Participants
    ASA 1 | 40 | 39 | 79
    ASA 2 | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption in the Immediate Postoperative Period
Description: This data will be entered into the participants electronic medical record and collected from their chart once the participant has been discharged. The "immediate postoperative period" covers the participant's entire time in the outpatient surgery center after they have entered the recovery room postoperatively. The amount of time they remain in the outpatient surgery center postoperatively varies from a minimum of 1 hour to a maximum of 10 hours and an average of 4 hours.
Time Frame: Up to 10 hours
Measure: Mean (Standard Deviation); unit: morphine mg equivalents
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
morphine mg equivalents | 12.0 (11.9) | 14.4 (9.3)

2. Secondary Outcome: Pain Scores During Recovery
Description: Pain scores during recovery period through the first 24 hours of recovery, recorded upon arrival to recovery room, 1-hr post-op, 24-hrs post-op. This outcome reports lowest and highest pain score since discharge to 24 hour phone call. Pain scores are collected verbally on a scale of 0-10 where 10 is the most severe pain.
Time Frame: up to 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
score on a scale
  Lowest Score Upon Arrival to Recovery Room | 2.3 (2.1) | 3.0 (1.6)
  Highest Score Upon Arrival to Recovery Room | 4.8 (2.4) | 5.5 (2.0)
  1 hour post-op | 3.4 (1.9) | 3.8 (1.6)
  24 hours post-op | 2.4 (1.8) | 2.6 (1.7)

3. Secondary Outcome: Number of Participants Who Received Medication for Nausea
Description: Number of participant who received medication for nausea prior to discharge and after discharge, up to 24 hours post-op.
Time Frame: Up to 24 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
Participants
  Anti-Nausea Medication Before Discharge | 8 | 7
  Anti-Nausea Medication after Discharge | 6 | 3

4. Secondary Outcome: Post-Operative Incidence of Nausea
Description: Incidence of nausea as recorded in the electronic medical record (EMR) in the recovery room through the first 24-hrs post-op.
Time Frame: Up to 24 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
Participants
  Nausea Post op to discharge | 16 | 12
  Nausea - discharge to 24 hour | 24 | 23

5. Secondary Outcome: Post-Operative Nausea Scores
Description: Nausea scores will be collected in post-operative recovery and 24 hours later (via phone). The participant will be asked to rate their nausea on a scale of 0 (no nausea) - 10 (worst possible).
Time Frame: Up to 24 hours following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
score on a scale
  Post Operative (recovery room) | 1.2 (2.3) | 0.7 (1.7)
  24 hours post-op | 2.2 (3.0) | 1.6 (2.7)

6. Secondary Outcome: Incidence of Post-Operative Pruritus
Description: Pruritus in recovery and through the first 24 hours post-op.
Time Frame: Up to 24 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
Participants
  Number of patients with pruritis OR to discharge | 8 | 10
  Number of patients with pruritis discharge to 24 h | 13 | 19

7. Secondary Outcome: Post-Operative Pruritis Score
Description: Participants will be asked to rate their pruritis on a scale of 0 (no itching) - 10 (worst itchiness) while in post-op recovery room and then at 24 hours post-op via phone call.
Time Frame: Up to 24 hours following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
score on a scale
  Post Operative (recovery room) | 0.4 (1.0) | 0.7 (1.7)
  24 hours post-op | 0.7 (1.4) | 1.2 (2.1)

8. Secondary Outcome: Sedation Scale
Description: Sedation scale measured in recovery room, 1-hr post op, and 24 hrs op. The Sedation Scale is scored from 0-10 where 0 = normal, no sleepier than average, 10 = sleepy, hard to stay awake.
Time Frame: Up to 24 hours following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
score on a scale
  1 hour post-op in Recovery Room | 5.0 (2.3) | 4.6 (2.2)
  24 hours post-op | 4.2 (3.0) | 4.3 (2.8)

9. Secondary Outcome: Impact of Block Characteristics on Pain Control
Time Frame: Up to 24 hours following surgery
Population: This data was not collected. All participants had a femoral nerve block. The quality of this block was not assessed.
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Intraoperative Medication Use: Ketorolac and Lidocaine
Description: All participants received standard induction medications.
Time Frame: From induction until arrival in post anesthesia care unit.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
mg
  Intraoperative Ketorolac | 15.0 (4.1) | 14.7 (4.5)
  Intraoperative Lidocaine | 71.5 (28.4) | 65.6 (36.9)

11. Secondary Outcome: Intraoperative Medication Use: Fentanyl
Description: All participants received standard induction medications.
Time Frame: From induction until arrival in post anesthesia care unit.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
mcg | 125 (64.4) | 128 (81.8)

12. Secondary Outcome: Number of Participants With Complications From the Procedure
Time Frame: Up to 24 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
Participants | 0 | 0

13. Secondary Outcome: Time to Discharge
Description: Time to discharge from the recovery room (Phase I recovery) and the outpatient surgery center (Phase II recovery).
Time Frame: Up to 24 hours following surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
Number analyzed (Participants) | 55 | 57
minutes
  Discharge from Recovery Room | 64.8 (17.7) | 61.4 (19.5)
  Discharge from Outpatient Center | 132.1 (64.2) | 123.6 (48.6)

ADVERSE EVENTS:
Time Frame: up to 24 hours post-op
Arm/Group | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine | Placebo Pills and Injectables
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/57
Other Adverse Events (participants affected / at risk) | 0/55 | 3/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multimodal:Acetaminophen, Gabapentin, Ketamine, Bupivacaine (N=55) | Placebo Pills and Injectables (N=57)
Light Headed After Surgery (Surgical and medical procedures) | 0 | 1
Vivid Dreams (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT01868425/Prot_SAP_001.pdf